CLINICAL TRIAL: NCT02367079
Title: Diathermy Compared With Sham Diathermy in Doms Management
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: 1 day data collection
Sponsor: Studi Fisioterapici di Montagna (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Treatment
Other Study IDs: StudiFM
Record Dates: First submitted 2015-01-21; First posted 2015-02-20 (Estimated); Last update posted 2015-02-20 (Estimated); Status verified 2015-02

CONDITIONS: Musculoskeletal Diseases
MeSH Terms: conditions — Musculoskeletal Diseases | interventions — Diathermy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Switched on diathermy (Active Comparator): Switched on diathermy was used on DOMS compared to sham diathermy
  Interventions: Device: Diathermy
- Switched OFF diathermy (Sham Comparator): Switched OFF diathermy was used on DOMS compared to REAL diathermy
  Interventions: Device: Diathermy

INTERVENTIONS:
Device: Diathermy — Sham diathermy vs switched on diathermy effect on pain where assessed

SUMMARY:
To investigate the effect of hand massage, switched on diathermy or sham/switched off diathermy on DOMS in a group of athletes suffering DOMS after a ski mountaineering race.

DETAILED DESCRIPTION:
This study examine DOMS in athletes following a ski mountaineering race, pain measured with numbering pain rating scale NPRS and perceived global improvement (PGIC) after treatment have been measured after a massage treatment, a diathermy treatment and a sham diathermy treatment.

ELIGIBILITY:
Inclusion Criteria:

- Healthy patients who complaints about D.O.M.S. after a skimountaneering race

Exclusion Criteria:

- Patient who complain of pathology such trauma or declaring consuming drugs for pain management where excluded from the study.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2014-04; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Numering pain rating scale | Day 1
  Numering pain rating scale was assessed pre e post treatment

CONTACTS AND LOCATIONS:
Overall Officials: LORENZO VISCONTI, Bsc, Principal Investigator — Studi Fisioterapici di Montagna
Locations (1):
- Studi fisioterapici di Montagna, Aosta, Aosta, Italy